CLINICAL TRIAL: NCT04838080
Title: Phase 1 Study for the Determination of Safety and Immunogenicity of Different Strengths of Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine, Given Twice Intramuscularly to Healthy Volunteers, in a Placebo Controlled Study Design.
Brief Title: Safety and Immunogenicity of the Inactivated Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine Compared to Placebo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocak Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALP-2020-FZ-01-PK-537-2
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19; Vaccine; Inactive; Phase 1
MeSH Terms: conditions — COVID-19; Sedentary Behavior | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose vaccine (Experimental): Inactivated COVID-19 Vaccine 4 µg/0.5 ml
  Interventions: Biological: Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine 4 µg/0.5 ml Vaccine
- High Dose Vaccine (Experimental): Inactivated COVID-19 Vaccine 6 µg/0.5 ml
  Interventions: Biological: Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine 6 µg/0.5 ml Vaccine
- Placebo (Placebo Comparator): 0.9 % NaCl
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine 4 µg/0.5 ml Vaccine — Two applications on Days 0 and 21
  Arms: Low dose vaccine
Biological: Koçak-19 Inaktif Adjuvanlı COVID-19 Vaccine 6 µg/0.5 ml Vaccine — Two applications on Days 0 and 21
  Arms: High Dose Vaccine
Biological: Placebo — Two applications on Days 0 and 21
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the safety and immunogenicity of two different strengths (4 µg and 6 µg) of an inactivated COVID-19 Vaccine compared to placebo so that to demonstrate the safety and efficacy in prophylaxis of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* healthy Caucasian origin
* male or female
* age between 18 and 55 years
* accepting not to participate in another COVID-19 vaccine study until the end of the study
* volunteers who do not plan to get a child in the next one year; the volunteer and the partner should use a reliable form of contraception (abstinence, condom, birth control implant, birth control pills used or IUD used by the partner) during the study for at least 1 year
* female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months) must agree to be heterosexually inactive through 12 months after the first vaccination OR agree to consistently use any of the described methods of contraception from through 12 months after the first vaccination.
* male subjects agree to refrain from sperm donation from the time of first vaccination until 3 months after last vaccination
* participants must refrain from blood or plasma donation from the time of first vaccination until 3 months after last vaccination
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* life style and habits (consumption of alcohol, nicotine, coffee, tea, coke, special diet, drug abuse) should be normal/acceptable
* body temperature, pulse rate, blood pressure, respiratory rate and 12 lead ECG should be normal/acceptable.
* physical examination (general state and abnormal findings per system: endocrine/metabolic, allergies, drug sensitivities, head, neck, eyes, ears, nose, throat, cardiovascular, respiratory, gastrointestinal, hepatic/biliary, urogenital, musculoskeletal, Lymph nodes, skin, and neurological/psychiatric) should be normal/acceptable
* laboratory examination (blood/serum examination: sodium, potassium, calcium, chloride, total protein, albumin, glucose, creatinine, BUN, uric acid, total bilirubin, direct and indirect bilirubin, lipid panel (total cholesterol, triglyceride, HDL, LDL), AST, ALT, GGT, ALP, haemoglobin, haematocrit, erythrocytes, Leukocytes, platelet count, prothrombin time (PT) and activated partial thromboplastin time (aPTT); HBsAg, HIV-Ab, HCV-Ab; urine examination: urine color, appearance, specific gravity, pH, protein, glucose, ketones, blood, leukocytes, bilirubin, urobilinogen, nitrites and sediment if erythrocytes or leucocytes are out of the limits ) should be normal/acceptable.
* antiSARS CoV 2 total antibody (including COVID-19 IgG and/or IgM) negative in serum.
* drug screening negative (amphetamines, cannabinoids, benzodiazepines, cocaine, opioids, barbiturates)
* normal body weight in relation to height and age according to
* BMI = weight(kg) / height (m)2 (accepted range 18.5 and 30 kg/m2)
* Informed consent given in written form according to section 15.3.
* agree not to participate in another vaccine clinical trial until the end of the study.
* agree to remain in the study area for the entire duration of the study.

Exclusion Criteria:

* women with a positive blood (β-HCG) pregnancy test
* lactating women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.
* positive real time RT-PCR COVID-19 test.
* leukemia or neoplasm in history.
* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 30 days before the first dose
* presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, haematological, gastrointestinal, neurological, psychiatric or other major diseases;
* disruption of platelets or other blood clotting disorders, which may cause contraindications to intramuscular administration
* clinically significant illness within 4 weeks before the start of the study. Especially any acute or chronic illness seizures.
* any regular intake or administration of any prescribed systemic or topical medication within 2 weeks prior to the start of the study; in the case of intake or administration of any prescribed systemic or topical medication within 4 weeks before the start of the study because of an insignificant illness, this should be stated in the CRF.
* intake or administration of OTC medication (including herbal remedies) which may have an effect on the study according to the investigator within 2 weeks prior to the start of the study
* volunteers who received antiviral drugs, immunoglobulins or blood transfusions or any other investigational drug within 4 weeks prior to the first study product administration
* concomitant intake or administration of any systemic or topical drugs (including herbal remedies) on the application days
* treatment with any investigational drug (i.e., drug not yet approved) in the last 4 weeks before beginning of the trial
* medication with drugs known to alter organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 1 month (4 weeks)
* donation of blood or plasma more than 450 ml within the last 2 months (8 weeks) or any amount within the last month (4 weeks)
* supine blood pressure, after resting for 5 min, higher than 140/90 or lower than 100/60 mmHg
* supine pulse rate, after resting for 5 min, outside the range of 50 - 100 beats/min
* supine respiratory rate, after resting for 5 min, outside the range of 15 - 18 breathings / min
* any clinically significant abnormality of the ECG (12 leads) recorded in rest
* laboratory values (appendix 5) outside normal range with clinical relevance at entry examination
* alcohol abuse i.e. regular use of more than 2 units of alcohol per day or a history of alcoholism or drug/chemical abuse (one unit of alcohol equals ½ l of beer, 200 ml wine or 50 ml of spirits) or recovered alcoholics
* caffeine abuse i.e. regular use of more than 750 mg/day caffeine
* alcoholic or methylxanthine-containing beverages or foods (coffee, tea, coke, chocolate) and fruit-juice from 24 hours prior to each application until the end of hospitalization
* grapefruit products from 7 days prior to the first application until the end of hospitalization
* smoking of more than 10 cigarettes or equivalent per day, no smoking allowed during hospitalization in the clinical unit
* vegetarian or any special diet due to any reason
* knowledge to have any type of parenterally transmitted hepatitis or carrier of the HBsAg (HBsAg test positive)
* HIV-Ab test positive
* Test on anti-HCV antibodies positive
* positive drug screen or history of drug abuse (amphetamines, cannabinoids, benzodiazepines, cocaine, opioids, barbiturates)
* legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study
* evidence of an uncooperative attitude.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women
Enrollment: 38 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-20 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From day 0 until the end of follow up period (6 months)
  Questioning adverse events and examination of laboratory safety data

SECONDARY OUTCOMES:
Serum immunoglobulin G (IgG) antibody levels | From screening until the end of follow up period (6 months)
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s)
Neutralizing antibodies | From screening until the end of follow up period (6 months)
  Measurement of SARS-CoV-2-specific neutralizing antibodies
Blood levels of cytokines | From screening until the end of follow up period
  TNF-alpha, IFN-γ, IL-2, IL-4, IL-5 and IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Aydin Erenmemisoglu, Prof., Study Director — Legal representative; Turgay Celik, Prof., Principal Investigator — Principal Investigator
Locations (1):
- Yeditepe AR-GE ve Analiz Merkezi İyi Klinik Uygulamaları Merkezi (Center for GCP), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No